CLINICAL TRIAL: NCT03730012
Title: Phase 1/2 Study of ASP2215 (Gilteritinib) Combined With Atezolizumab in Patients With Relapsed or Treatment Refractory FLT3 Mutated Acute Myeloid Leukemia (AML)
Brief Title: A Study of ASP2215 (Gilteritinib) Combined With Atezolizumab in Patients With Relapsed or Treatment Refractory FMS-like Tyrosine Kinase (FLT3) Mutated Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-1101
Expanded Access: NCT03070093 (Approved for marketing)
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Results first posted 2022-06-24 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Myeloid Leukemia With FMS-like Tyrosine Kinase (FLT3) Mutation
Keywords: AML; gilteritinib; ASP2215; Acute Myeloid Leukemia; FLT3
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gilteritinib 120 mg + Atezolizumab 420 mg (Experimental): Participants received 120 milligrams (mg) giltertinib (3 tablets of 40 mg) orally, once a day in continuous 28-day cycles in combination with atezolizumab 420 mg adminstered by intravenous infusion (over 60 minutes) once every 2 weeks of 28-day cycle until the participant no longer received clinical benefit from therapy, unacceptable toxicity occurred or the participant met a treatment discontinuation criterion (Maximum treatment duration was 535 days for gilteritinib and 112 days for atezolizumab).
  Interventions: Drug: gilteritinib; Drug: atezolizumab
- Gilteritinib 120 mg + Atezolizumab 840 mg (Experimental): Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day in continuous 28-day cycles in combination with atezolizumab 840 mg administered by intravenous infusion (over 60 minutes) once every 2 weeks of 28-day cycle until the participant no longer received clinical benefit from therapy, unacceptable toxicity occurred or the participant met a treatment discontinuation criterion (Maximum treatment duration was 126 days for gilteritinib and 70 days for atezolizumab).
  Interventions: Drug: gilteritinib; Drug: atezolizumab

INTERVENTIONS:
Drug: gilteritinib — Oral tablet
  Other Names: ASP2215
Drug: atezolizumab — Intravenous infusion

SUMMARY:
The purpose of this study was to determine the safety and tolerability of gilteritinib given in combination with atezolizumab in participants with relapsed or treatment refractory FMS-like tyrosine kinase 3 (FLT3) mutated AML and to determine the composite complete remission (CRc) rate for participants who either discontinued the study or completed 2 cycles of gilteritinib given in combination with atezolizumab.

This study also evaluated pharmacokinetics (PK), response to treatment, remission and survival. Adverse events (AEs), clinical laboratory results, vital signs, electrocardiograms (ECGs), and Eastern Cooperative Oncology Group (ECOG) performance status scores were also assessed.

DETAILED DESCRIPTION:
This study was planned to have 2 phases:

Phase 1:

The phase 1 portion of this study was to establish the recommended phase 2 dose (RP2D) of gilteritinib given in combination with atezolizumab.

Phase 2:

The phase 2 portion of the study was to treat participants with gilteritinib and atezolizumab at the RP2D and was to be enrolled in two stages. The first stage was to evaluate the remission rate and if a minimum rate was to be achieved, a second stage of enrollment was to be continued.

ELIGIBILITY:
Inclusion Criteria:

* Subject is considered an adult according to local regulation at the time of signing informed consent form (ICF).
* Subject has defined AML by the World Health Organization (WHO) criteria (2017) and fulfills one of the following:

  * Refractory to at least 1 cycle of induction chemotherapy
  * Relapsed after achieving remission with a prior therapy
* Subject is positive for FLT3 mutation in bone marrow or blood after completion of the subject's last interventional treatment.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 at screening.
* Subject must meet the following criteria as indicated on the clinical laboratory tests:

  * Serum Aspartate aminotransferase (AST) and Alanine Aminotransferease (ALT) ≤ 2.5 x upper limit of normal (ULN)
  * Serum total bilirubin (TBL) ≤ 1.5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or an estimated glomerular filtration rate of > 50 mL/min as calculated by the Modification of Diet in Renal Disease equation.
* Subject is suitable for oral administration of study drug.
* A female subject is eligible to participate if she is not pregnant and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 180 days after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for at least 180 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for at least 180 days after the final study drug administration.
* A male subject must not donate sperm starting at screening and throughout the treatment period, and for at least 120 days after the final study drug administration.
* A male subject with female partner(s) of child-bearing potential must agree to use contraception during the treatment period, and for at least 120 days after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the treatment period, and for 120 days after the final study drug administration.
* Subject agrees not to participate in another investigational study while on treatment.

Exclusion Criteria:

* Subject was diagnosed as acute promyelocytic leukemia.
* Subject has BCR-ABL-positive leukemia (chronic myelogenous leukemia in blast crisis).
* Subject has AML secondary to prior chemotherapy for other neoplasms (except for myelodysplastic syndrome).
* Subject has clinically active central nervous system leukemia.
* Subject has uncontrolled or significant cardiovascular disease, including:

  * A myocardial infarction within 12 months
  * Uncontrolled angina within 6 months
  * History of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, torsades de pointes) or any history of arrhythmia
  * Uncontrolled hypertension
* Subject has baseline left ventricular ejection fraction that is ≥ 45%.
* Subject has mean triplicate Fridericia-corrected QT interval (QTcF) > 450 ms at Screening based on central reading.
* Subject has congenital or acquired Long QT Syndrome at screening.
* Subject has hypokalemia and/or hypomagnesemia at screening.
* Subject has been diagnosed with another malignancy that requires concurrent treatment or hepatic malignancy regardless of the need for treatment.
* Subject has clinically significant coagulation abnormality unless secondary to AML.
* Subject is receiving or plans to receive concomitant chemotherapy or immunotherapy.
* Subject has had major surgery within 4 weeks prior to the first study dose.
* Subject has radiation therapy within 4 weeks prior to the first study dose.
* Subject requires treatment with concomitant drugs that are strong inducers of Cytochrome P450 (CYP3A).
* Subject has known pulmonary disease with diffusion capacity of lung for carbon monoxide ≤ 65%, forced expiratory volume in the first second (FEV1) ≤ 65%, dyspnea at rest or requiring oxygen or any pleural neoplasm.
* Subject with systemic fungal, bacterial, viral or other uncontrolled infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment. Subject needs to be off pressors and have negative blood cultures for 48 hours.
* Subject has not recovered from any prior therapy related toxicities.
* Subject is known to have human immunodeficiency virus infection.
* Subject has active hepatitis B or C or other active hepatic disorder.
* Subject has previously been treated with gilteritinib, quizartinib or crenolanib (will only apply to subjects enrolled in the phase 2 portion of the study).
* Subject has active clinically significant graft-versus-host disease (GVHD) or is on treatment with systemic corticosteroids for GVHD.
* Subject has relapsed after allogeneic hematopoietic stem cell transplant (HCST).
* Subject has an active autoimmune disorder that makes the subject unsuitable for study treatment or participation.
* Subject has any condition that makes the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development
Locations (12):
- United States (12):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Roswell Park Cancer Institute (RPCI), Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - The Ohio State University Comprehensive Cancer Center (OSUCCC), Columbus, Ohio
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Simmons Comprehensive Cancer Center, Dallas, Texas
  - University of Texas MD Anderson, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://www.clinicaltrials.astellas.com/study/?pid=2215-CL-1101
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14793&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was planned for two phases, dose-escalation (phase 1) and dose expansion (phase 2). Sponsor decided not to open the phase 2 extension part of the study after completion of phase 1 dose escalation part.
Pre-assignment Details: Participants with relapsed or treatment refractory FMS-like tyrosine kinase 3 (FLT3) mutated acute myeloid leukemia (AML) were enrolled in this study.
Groups:
- Gilteritinib 120 mg + Atezolizumab 420 mg: Participants received 120 mg (milligrams) giltertinib (3 tablets of 40 mg) orally, once a day in continuous 28-day cycles in combination with atezolizumab 420 mg adminstered by intravenous infusion (over 60 minutes) once every 2 weeks of 28-day cycle until the participant no longer received clinical benefit from therapy, unacceptable toxicity occurred or the participant met a treatment discontinuation criterion (Maximum treatment duration was 535 days for gilteritinib and 112 days for atezolizumab).
- Gilteritinib 120 mg + Atezolizumab 840 mg: Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day in continuous 28-day cycles in combination with atezolizumab 840 mg adminstered by intravenous infusion (over 60 minutes) once every 2 weeks of 28-day cycle until the participant no longer received clinical benefit from therapy, unacceptable toxicity occurred or the participant met a treatment discontinuation criterion (Maximum treatment duration was 126 days for gilteritinib and 70 days for atezolizumab).
Period: Overall Study
Arm/Group | Gilteritinib 120 mg + Atezolizumab 420 mg | Gilteritinib 120 mg + Atezolizumab 840 mg
Started | 3 | 8
Completed | 0 | 0
Not Completed | 3 | 8
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 1 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Miscellaneous | 2 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who took at least 1 dose of study drug (gilteritinib or atezolizumab).
Groups:
- Gilteritinib 120 mg + Atezolizumab 420 mg: Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day in continuous 28-day cycles in combination with atezolizumab 420 mg adminstered by intravenous infusion (over 60 minutes) once every 2 weeks of 28-day cycle until the participant no longer received clinical benefit from therapy, unacceptable toxicity occurred or the participant met a treatment discontinuation criterion (Maximum treatment duration was 535 days for gilteritinib and 112 days for atezolizumab).
- Total: Total of all reporting groups
Arm/Group | Gilteritinib 120 mg + Atezolizumab 420 mg | Gilteritinib 120 mg + Atezolizumab 840 mg | Total
Number analyzed (Participants) | 3 | 8 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (8.7) | 64.8 (20.8) | 68.4 (18.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 8 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT)
Description: DLTs were defined as:
  * Confirmed Hy's Law case
  * Any Grade ≥ 3 non-hematologic or extramedullary toxicity with the following exceptions:
    * Anorexia or fatigue
    * Grade 3 nausea and/or vomiting if participant did not require tube feeding or total parenteral nutrition, or diarrhea if the events did not require or prolong hospitalization that could be managed to grade ≤ 2 with standard antiemetic or antidiarrheal medications used at prescribed dose within 7 days of onset.
    * Grade 3 mucositis that resolved to Grade ≤ 2 within 7 days of onset
    * Grade 3 fever with neutropenia, with or without infection
    * Grade 3 infection
    * Grade 3 infusion-related toxicity, if successfully managed and resolved within 72 hours.
Time Frame: Day 1 up to 28 days
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Gilteritinib 120 mg + Atezolizumab 420 mg | Gilteritinib 120 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 8
Participants | 0 | 2

2. Secondary Outcome: Composite Complete Remission (CRc) Rate
Description: CRc was defined as rate of all complete and incomplete remissions i.e. CR + CR with incomplete platelet recovery (CRp) + CR with incomplete hematological recover (CRi).
  Participants were classified as:
  CR if they achieved morphologic leukemia-free state & their bone marrow was regenerating normal hematopoietic cells. If they had absolute neutrophil count (ANC) > 1 × 10^9/L, platelet count ≥ 100 × 10^9/L, normal marrow differential < 5% blasts, & were red blood cell (RBC) and platelet transfusion independent (defined as 1 week without RBC transfusion and platelet transfusion prior to disease assessment). There was also no evidence of extramedullary leukemia.
  CRp if they achieved CR with incomplete platelet recovery (< 100 × 10^9/L). CRi if they achieved CR with incomplete hematological recovery with residual neutropenia < 1 × 10^9/L, with or without complete platelet recovery. RBC and platelet transfusion independence was not required.
  Percentage of participants with CRc was reported.
Time Frame: From the date of first dose up to end of treatment (Maximum treatment duration was 535 days for gilteritinib and 112 days for atezolizumab)
Population: The full analysis set (FAS) consisted of all participants who were enrolled in the study and took at least 1 dose of study drug (gilteritinib or atezolizumab).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gilteritinib 120 mg + Atezolizumab 420 mg | Gilteritinib 120 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 8
Percentage of participants | 33.3 [0.8 to 90.6] | 12.5 [0.3 to 52.7]

3. Secondary Outcome: Plasma Ctrough Concentration of Gilteritinib
Description: Plasma Ctrough concentrations of gilteritinib was reported. One cycle = 28 days.
  C= cycle, D=day
Time Frame: Pre-dose on C1D1, C1D8, C1D15, C2D1,C2D15, C3D1, C3D15, C4D1, C4D15, C5D1, C5D15, C6D1, C6D15
Population: The pharmacokinetic analysis set (PKAS) consisted of the administered population for which sufficient plasma concentration data was available to facilitate derivation of at least 1 PK parameter and for whom at least 1 plasma concentration datum was available and both the date and time of dosing on the day of PK sampling and the date and time of sampling were known. Participants with available data at specified time point were included.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Gilteritinib 120 mg + Atezolizumab 420 mg | Gilteritinib 120 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 7
Nanogram per milliliter
  Pre-dose C1D1 | NA (NA) — Concentrations below the limit of quantification (10 nanogram per milliliter) | NA (NA) — Concentrations below the limit of quantification (10 nanogram per milliliter)
  Pre-dose C1D8 | 355 (240) | 302 (155)
  Pre-dose C1D15: number analyzed (Participants) | 3 | 4
  Pre-dose C1D15 | 483 (272) | 553 (436)
  Pre-dose C2D1: number analyzed (Participants) | 1 | 3
  Pre-dose C2D1 | 228 | 422 (328)
  Pre-dose C2D15: number analyzed (Participants) | 0 | 1
  Pre-dose C2D15 |  | 83.3
  Pre-dose C3D1: number analyzed (Participants) | 0 | 1
  Pre-dose C3D1 |  | 62.1
  Pre-dose C3D15: number analyzed (Participants) | 0 | 1
  Pre-dose C3D15 |  | 75.2
  Pre-dose C4D1: number analyzed (Participants) | 0 | 0
  Pre-dose C4D15: number analyzed (Participants) | 0 | 0
  Pre-dose C5D1: number analyzed (Participants) | 0 | 0
  Pre-dose C5D15: number analyzed (Participants) | 0 | 0
  Pre-dose C6D1: number analyzed (Participants) | 0 | 0
  Pre-dose C6D15: number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Complete Remission (CR) Rate
Description: Participants were classified as CR if they achieved a morphologic leukemia-free state and their bone marrow was regenerating normal hematopoietic cells. In addition, these participants had ANC > 1 × 10^9/L, platelet count ≥ 100 × 10^9/L, normal marrow differential with < 5% blasts, and were RBC and platelet transfusion independent (defined as 1 week without RBC transfusion and 1 week without platelet transfusion prior to disease assessment). There was also no evidence of extramedullary leukemia. CR rate was defined as the number of participants with CR divided by the number of participants in the analysis population. Percentage of participants with CR was reported.
Time Frame: as for outcome 2
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gilteritinib 120 mg + Atezolizumab 420 mg | Gilteritinib 120 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 8
Percentage of participants | 33.3 [0.8 to 90.6] | 0 [0 to 0]

5. Secondary Outcome: Complete Remission With Partial Hematologic Recovery (CRh) Rate
Description: Participants were classified as CRh if they achieved CR with ANC level of > 0.5 × 10^9/L and platelet count of > 50 × 10^9/L. CRh rate was defined as the number of participants with CRh divided by the number of participants in the analysis population.
  Participants were classified as CR if they achieved a morphologic leukemia-free state and their bone marrow was regenerating normal hematopoietic cells. In addition, these participants had ANC > 1 × 10^9/L, platelet count ≥ 100 × 10^9/L, normal marrow differential with < 5% blasts, and were RBC and platelet transfusion independent (defined as 1 week without RBC transfusion and 1 week without platelet transfusion prior to disease assessment). There was also no evidence of extramedullary leukemia. Percentage of participants with CRh was reported.
Time Frame: as for outcome 2
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gilteritinib 120 mg + Atezolizumab 420 mg | Gilteritinib 120 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 8
Percentage of participants | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Best Response Rate
Description: Best response was defined as the best-measured response (CR, CRp, CRi or PR) post-treatment. Best response rate was defined as the number of participants with CR or CRp or CRi or PR divided by the number of participants in the analysis population (i.e., CR+ CRp + CRi + PR). Participants with unknown or missing response, or who provide no information on response at the end of study will be treated as non-responders and will be included in the denominator when calculating rates. CR, CRp and CRi were described in outcome measure 2#. Participants were classified as PR if their bone marrow was regenerating normal hematopoietic cells with evidence of peripheral recovery with no (or only a few regenerating) circulating blasts and a decrease of at least 50% in the percentage of blasts in the bone marrow aspirate/biopsy, with the total marrow blasts between 5% and 25%. Percentage of participants with best response was reported.
Time Frame: as for outcome 2
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gilteritinib 120 mg + Atezolizumab 420 mg | Gilteritinib 120 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 8
Percentage of participants | 33.3 [0.8 to 90.6] | 25 [3.2 to 65.1]

7. Secondary Outcome: Duration of Remission (DoR)
Description: DoR: duration of CRc, CR, CRi, CRp & response (CRc + PR). Duration of CRc/CR/CRi/CRp: time from date of first CRc/CR/CRi/CRp until date of documented relapse for participants who achieved CRc/CR/CRi/CRp. Duration of response: time from date of either first CRc or PR until date of documented relapse of any type for participants who achieved CRc or PR. CRc, CR, CRi, CRp were described in outcome measure #2 & PR was described in outcome measure #6. Relapse after CR, CRp or CRi: reappearance of leukemic blasts in peripheral blood or ≥ 5% blasts in bone marrow aspirate/biopsy not attributable to any other cause or reappearance or new appearance of extramedullary leukemia. Relapse after PR: reappearance of significant numbers of peripheral blasts & an increase in the percentage of blasts in the bone marrow aspirate/biopsy to > 25% not attributable to any other cause or reappearance or new appearance of extramedullary leukemia. Analysis was performed using Kaplan-Meier estimates.
Time Frame: From date of first response until the date of documented relapse (Maximum treatment duration was 535 days for gilteritinib and 112 days for atezolizumab)
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Gilteritinib 120 mg + Atezolizumab 420 mg | Gilteritinib 120 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 8
Days | NA [NA to NA] — Median, upper and lower limit of 95% CI were not estimable due to low number of events. | NA [31.0 to NA] — Median and upper limit of 95% CI were not estimable due to low number of events.

8. Secondary Outcome: Event Free Survival (EFS)
Description: EFS was defined as time from date of first dose until date of documented relapse from CR, CRp or CRi, treatment failure or death from any cause, whichever occurred first. CRc, CR, CRi, CRp were described in Outcome measure #2. For a participant with none of these events, EFS was censored at date of last disease assessment. Relapse after CR, CRp or CRi was defined as reappearance of leukemic blasts in peripheral blood or ≥ 5% blasts in bone marrow aspirate/biopsy not attributable to any other cause or reappearance or new appearance of extramedullary leukemia. Relapse after PR was defined with reappearance of significant numbers of peripheral blasts & an increase in the percentage of blasts in the bone marrow aspirate/biopsy to > 25% not attributable to any other cause or reappearance or new appearance of extramedullary leukemia. Treatment failure was defined as lack of CR, CRp or CRi, & was determined at the end of treatment (EoT). Analysis was performed using Kaplan-Meier estimates.
Time Frame: From the date of first dose until the date of documented relapse from CR, CRp or CRi, treatment failure or death from any cause, whichever occurred first (Maximum treatment duration was 535 days for gilteritinib and 112 days for atezolizumab)
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Gilteritinib 120 mg + Atezolizumab 420 mg | Gilteritinib 120 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 8
Days | 175.00 [71.00 to NA] — Upper limit of 95% CI was not estimable due to low number of events. | 52.50 [2.00 to 58.00]

9. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose until the date of death from any cause. For a participant who was not known to have died by the end of study follow-up, overall survival was censored at the date of last contact. Analysis was performed using Kaplan-Meier estimates.
Time Frame: From the date of first dose until the date of death from any cause (Maximum treatment duration was 535 days for gilteritinib and 112 days for atezolizumab)
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Gilteritinib 120 mg + Atezolizumab 840 mg | Gilteritinib 120 mg + Atezolizumab 420 mg
Number analyzed (Participants) | 3 | 8
Days | 175.00 [111.00 to NA] — Upper limit of 95% CI was not estimable due to low number of events. | NA [51.00 to NA] — Median and upper limit of 95% CI was not estimable due to low number of events.

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: An AE was any untoward medical occurrence in a participant administered study drug, & which did not necessarily have to have a causal relationship with this treatment. Abnormalities was defined as AE only if met 1 of the criteria:Induced clinical signs/symptoms, required active intervention, required interruption or discontinuation of ST, abnormality or investigational value was clinically significant. Serious AE:resulted in death, was life threatening, persistent or significant disability/incapacity or substantial disruption of ability to conduct normal life functions, congenital anomaly/birth defect, required hospitalization or prolongation of hospitalization, other medically important events. Any AE recorded on treatment including within 30 days from last study treatment was classified as treatment-emergent AE (TEAE). Grades(Gr) based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE) (Gr 1=mild, Gr 2=moderate, Gr 3 =severe, Gr 4 =life threatening, Gr 5 =death).
Time Frame: Baseline to 30 days after last study treatment (Maximum treatment duration was 535 days for gilteritinib and 112 days for atezolizumab)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Gilteritinib 120 mg + Atezolizumab 420 mg | Gilteritinib 120 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 8
Participants
  TEAE | 3 | 8
  Drug-Related Adverse Events | 3 | 7
  TEAE leading to Deaths | 1 | 2
  Drug-related TEAE Leading to Deaths | 0 | 0
  Serious Adverse Events | 3 | 7
  Drug-Related Serious Adverse Events | 3 | 6
  Adverse Events Leading to Withdrawal of Treatment | 2 | 6
  Drug-Related Adverse Events Leading to Withdrawal of Treatment | 1 | 5
  Grade 3 or Higher TEAE | 3 | 8
  Treatment Emergent Deaths | 1 | 2

11. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Score
Description: ECOG performance status was measured on an 6 point scale. 0-Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. Dead.
Time Frame: Baseline and end of treatment (EoT) (Maximum treatment duration was 535 days for gilteritinib and 112 days for atezolizumab)
Population: Safety population with available data at specified timepoint
Measure: Number; unit: Participants
Arm/Group | Gilteritinib 120 mg + Atezolizumab 420 mg | Gilteritinib 120 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 8
Participants
  Baseline: Grade 0 | 0 | 3
  Baseline: Grade 1 | 3 | 4
  Baseline: Grade 2 | 0 | 1
  Baseline: Grade 3 | 0 | 0
  Baseline: Grade 4 | 0 | 0
  Baseline: Grade 5 | 0 | 0
  EoT: Grade 0: number analyzed (Participants) | 2 | 4
  EoT: Grade 0 | 0 | 1
  EoT: Grade 1: number analyzed (Participants) | 2 | 4
  EoT: Grade 1 | 1 | 1
  EoT: Grade 2: number analyzed (Participants) | 2 | 4
  EoT: Grade 2 | 0 | 1
  EoT: Grade 3: number analyzed (Participants) | 2 | 4
  EoT: Grade 3 | 1 | 1
  EoT: Grade 4: number analyzed (Participants) | 2 | 4
  EoT: Grade 4 | 0 | 0
  EoT: Grade 5: number analyzed (Participants) | 2 | 4
  EoT: Grade 5 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to 30 days after last study treatment (Maximum treatment duration was 535 days for giltertinib and 112 days for atezolizumab)
Arm/Group | Gilteritinib 120 mg + Atezolizumab 420 mg | Gilteritinib 120 mg + Atezolizumab 840 mg
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/8
Serious Adverse Events (participants affected / at risk) | 3/3 | 7/8
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilteritinib 120 mg + Atezolizumab 420 mg (N=3) | Gilteritinib 120 mg + Atezolizumab 840 mg (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (6) | 5 (6)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (3)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilteritinib 120 mg + Atezolizumab 420 mg (N=3) | Gilteritinib 120 mg + Atezolizumab 840 mg (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (4) | 2 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (3) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (4) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 4 (4)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ocular icterus (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridium bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (3)
Bacterial test positive (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood corticotrophin decreased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 3 (10)
Respiratory syncytial virus test positive (Investigations) | 1 (1) | 0 (0)
Serum ferritin increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 2 (5) | 1 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (6) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (3) | 0 (0)
Dizziness (Nervous system disorders) | 3 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (4)
Lethargy (Nervous system disorders) | 1 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Device leakage (Product Issues) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 2 (10) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT03730012/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT03730012/SAP_001.pdf